CLINICAL TRIAL: NCT02140359
Title: Enhancing Housing First Programs With a Social Network Substance Use Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, David Kennedy, Behavioral / Social Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R34DA034855 (NIH)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Alcohol Drinking; Drug Abuse; HIV
Keywords: homelessness; housing first; social networks; drug abuse; alcohol use; HIV
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group: Usual Care (No Intervention): Residents of a housing first permanent supporting housing program will be randomly assigned to this arm after screening and baseline assessments. They will meet with case managers according to the usual procedures for new residents and will be given a standard case manager interaction.
- Motivational Network Interview Recipients (Experimental): Residents of a housing first permanent supporting housing program will be randomly assigned to this arm after screening and baseline assessments. They will meet roughly every two weeks with a case manager and answer questions about their social network, will be shown visual feedback about their networks, and will participate in a motivational interview conducted by the case managers. The questions and visualizations will be facilitated by an electronic tool for presenting screens with questions, capturing responses, processing and visualizing social network data.
  Interventions: Behavioral: Motivational Network Interview

INTERVENTIONS:
Behavioral: Motivational Network Interview — Residents of a housing first permanent supporting housing program will be randomly assigned to this arm after screening and baseline assessments. They will meet roughly every two weeks with a case manager and answer questions about their social network, will be shown visual feedback about their networks, and will participate in a motivational interview conducted by the case managers. The questions and visualizations will be facilitated by an electronic tool for presenting screens with questions, capturing responses, processing and visualizing social network data.
  Arms: Motivational Network Interview Recipients

SUMMARY:
Housing First programs are promising approaches to transitioning substance using chronically homeless adults to affordable housing. However, Housing First programs need to provide support to residents to adjust to their changing social environments. The proposed project fulfills a critical gap by developing an electronic tool for a social network intervention using motivational interviewing techniques as well as results of a pilot test of the tool. The hypothesis to be tested is that Housing First residents who are given the intervention will be significantly more motivated to change their drinking, drug use, sexual risk behaviors, and social networks compared to controls receiving usual care.

DETAILED DESCRIPTION:
We propose a 3-year study to develop and pilot test a social network substance use and HIV-risk intervention for permanent supportive housing program residents in the Skid Row area of Los Angeles. The intervention will be developed for residents at the Skid Row Housing Trust (SRHT), one of the largest Housing First providers in Los Angeles. Housing First residents are not required to abstain from alcohol and drugs as a requirement of their residency. There is some evidence that providing housing rapidly to chronically homeless persons--along with support--helps to reduce substance use and HIV risk behaviors in the short term because homelessness is the primary cause of high-risk behavior. However, the evidence thus far is limited. One aspect that has not received much research attention is the needs of Housing First residents for support to transition their social networks while transitioning out of homeless into residency in a Housing First program. New residents are exposed to a wide range of potentially negative social influences while also having greater potential to reconnect with lost positive ties. This project will develop a social network intervention to residents of SRHT in order to increase their knowledge about their social networks and enhance their motivation to make necessary changes to improve their ability to reduce or continue to abstain from high-risk behavior. The intervention sessions will enhance the weekly support meetings that SRHT case workers already conduct with new residents during their first 6 months of residency. Case workers will be trained to deliver the 30-minute intervention sessions using a motivational interviewing style. The intervention will be developed so that case managers can deliver it with the aid of an electronic tablet device. The tablet will guide them in collecting information about the residents' social networks and then display several diagrams highlighting various aspects of the residents' networks. They will then use motivational interviewing techniques to guide residents to think about how their network currently functions, how they would like it to function, and what steps they can take to make changes necessary to achieve goals related to reducing their substance use and sexual risk behaviors. The intervention will be delivered by case managers across four sessions (at baseline and at two-week intervals). We anticipate that residents who participate in this intervention will develop new strategies in their interactions with their social networks that will facilitate a reduction in their high-risk behavior.

ELIGIBILITY:
Inclusion Criteria:

* New residents of Skid Row Housing Trust receiving permanent supportive housing

Exclusion Criteria:

* Age younger than 18
* Does not speak English
* Cognitively impaired either by identifying those having a diagnosis of dementia in the new resident intake interview or using the Short Blessed Scale Exam)
* Does not screen positive for past -year harmful AOD use using the AUDIT-C (a score > 4 for men and > 3 for women) and DAST (a score greater than 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Readiness to change alcohol and other drug use | Baseline and 13-14 weeks (post intervention)
  Measured with 12 item Readiness to Change Questionnaire (RTCQ) and a one item Contemplation Ladder
Readiness to change risky sexual behavior | Baseline and 13-14 weeks (post intervention)
  11 item Readiness to Change Risky Sexual Behavior (RTCQ-SB) scale a one item Contemplation Ladder
Self efficacy to change alcohol and other drug use | Baseline and 13-14 weeks (post intervention)
  Measured with two questionnaire items that assess the participant's importance and self-efficacy to stop alcohol and other drug use and 4 items from the Alcohol Abstinence Self-Efficacy Scale (AASE) which measure how confident participants feel in their ability to abstain from alcohol use when depressed, relaxed, craving substances, and offered alcohol.
Self efficacy to change risky sexual behavior | Baseline and 13-14 weeks (post intervention)
  Measured with 4 item Self-Efficacy to Use Condoms scale
Self-efficacy to change social networks | Baseline and 13-14 weeks (post intervention)
  Two item ladder scale item measuring importance and self-efficacy to change social networks.
Perceived Social Network support and approval/disapproval of alcohol, drug use, and risky sex. | Baseline and 13-14 weeks (after intervention)
  Measures of Perceived Social Support and ratings of network members on emotional closeness, drinking, drug use, safe-sex behavior, and approval/disapproval of high-risk behavior of social network members based on the Important People Drug and Alcohol Interview. Raw network data to provide measures will result from a personal network interview in which participants will name 20 network member and answer questions about each of them and their relationships with each other.

SECONDARY OUTCOMES:
Drug and Alcohol use | Baseline and 13-14 weeks (after intervention is completed)
  Assessed with a Timeline Followback calendar structured interview that measures alcohol and drug use through recall aided by a calendar. Participants will be asked quantity and intensity of drinking and drug use to calculate a quantity-frequency index for both drinking and drug use. Self-reports of non-use will be validated with a Oral Fluid Test.
HIV risk behavior | baseline and 13-14 weeks (after intervention completion)
  Survey items asking if the participant engaged in unprotected sex and concurrent sexual relationships overall and with particular partners in the past 90 days.
Change in social network composition and structure | baseline and 13-14 weeks (after intervention completion)
  Measures of network composition and structure will be constructed from raw network data. Raw network data result from a personal network interview in which participants will name 20 network member and answer questions about each of them and their relationships with each other.

OTHER OUTCOMES:
Satisfaction with Intervention | 13-14 weeks (after intervention)
  Administration of the Client Satisfaction Questionnaire (CSQ-8), an 8-item Likert-type measure of client feedback regarding services provided in a treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: David P Kennedy, PhD, Principal Investigator — RAND
Locations (2):
- United States (2):
  - Skid Row Housing Trust, Los Angeles, California
  - RAND Corporation, Santa Monica, California

REFERENCES:
- [Derived] Kennedy DP, Osilla KC, Hunter SB, Golinelli D, Maksabedian Hernandez E, Tucker JS. Restructuring personal networks with a Motivational Interviewing social network intervention to assist the transition out of homelessness: A randomized control pilot study. PLoS One. 2022 Jan 21;17(1):e0262210. doi: 10.1371/journal.pone.0262210. eCollection 2022. PMID 35061795
- [Derived] Osilla KC, Kennedy DP, Hunter SB, Maksabedian E. Feasibility of a computer-assisted social network motivational interviewing intervention for substance use and HIV risk behaviors for housing first residents. Addict Sci Clin Pract. 2016 Sep 7;11(1):14. doi: 10.1186/s13722-016-0061-x. PMID 27604543
- [Derived] Kennedy DP, Hunter SB, Chan Osilla K, Maksabedian E, Golinelli D, Tucker JS. A computer-assisted motivational social network intervention to reduce alcohol, drug and HIV risk behaviors among Housing First residents. Addict Sci Clin Pract. 2016 Mar 15;11(1):4. doi: 10.1186/s13722-016-0052-y. PMID 26979982